CLINICAL TRIAL: NCT00449748
Title: Evaluation of RAD001 as Therapy for Patients With Systemic Mastocytosis
Brief Title: Everolimus (RAD001) as Therapy for Patients With Systemic Mastocytosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2006-0759
Record Dates: First submitted 2007-03-19; First posted 2007-03-21 (Estimated); Results first posted 2011-04-29 (Estimated); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Systemic Mastocytosis
Keywords: Systemic Mastocytosis; RAD001
MeSH Terms: conditions — Mastocytosis, Systemic | interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- RAD001 (Experimental): Oral 10 mg daily for 30 days
  Interventions: Drug: RAD001 (Everolimus)

INTERVENTIONS:
Drug: RAD001 (Everolimus) — Oral RAD001 10 mg daily for 30 days

SUMMARY:
The goal of this clinical research study is to see if RAD001 can help to control the disease in patients with systemic mastocytosis (SM). The safety of this treatment will also be studied.

DETAILED DESCRIPTION:
RAD001 is designed to stop cancer cells from multiplying. It may also stop the growth of new blood vessels that help tumor growth, which may cause the tumor cells to die.

Before you can start treatment on this study, you will have "screening tests." These tests will help the doctor decide if you are eligible to take part in this study. They will be performed within 2 weeks before starting the study, unless listed otherwise. You will have a complete physical exam, including measurement of vital signs (blood pressure, heart rate, temperature, and breathing rate). Blood (about 2 tablespoons) will be drawn for routine tests. This routine blood draw will include a pregnancy test for women who are able to have children. To be eligible to take part in this study, the pregnancy test must be negative. You will need to "fast" for 6 hours before having these blood tests performed. This means you will not be able to have food or drink (except water) during this time.

Also as part of the screening tests, you will have an electrocardiogram (ECG)a test that measures the electrical activity of the heart). You will have a bone marrow biopsy and aspiration within 3 months of starting the study (or within 2 weeks of starting the study, if you have received treatment for SM). To collect a bone marrow biopsy/aspirate, an area of the hip bone is numbed with anesthetic, and a small amount of bone marrow and bone is withdrawn through a large needle. The bone marrow samples will be used not only to check the status of the disease, but also for a routine test to see if there is a mutation (change) in a certain gene. If your doctor feels it is necessary, you may need to have additional screening tests (such as a bone scan) to check the status of the disease.

If you are found to be eligible to take part in this study, you will receive your first supply of RAD001. You will take 1-2 pills of RAD001 by mouth once a day while you are on study. During the 3 hours before each dose of RAD001, you must eat no more than a light fat-free meal (such as a salad with no dressing, or a bowl of cereal with skim milk). You should also try to keep your dietary habits consistent before each dose. This means that you should eat at about the same time, and about the same amount of food each time.

Each "cycle" of RAD001 lasts 1 month. You will have study visits on Day 1 of Cycles 1, 2, and 3. At each visit, you will receive a new supply of RAD001. You will have a physical exam, including measurement of vital signs. You will be asked about any side effects you may have had. While you are on study, you must not take any additional medications (including over-the-counter products) without asking the study doctor first. At each study visit, you will be asked if you have taken any additional medications. You will also be asked if you have had any non-drug therapies or blood transfusions. Blood (about 2 tablespoons) will be drawn for routine tests. Like you did at screening, you will need to fast for 6 hours before having these blood tests performed.

Halfway through each cycle (at about the beginning of Week 3 of each cycle), blood will be drawn for routine tests. This will be about 2 tablespoons of blood each time. You will need to fast for 6 hours before having these blood tests performed. It is your choice whether to have these blood tests performed at M.D. Anderson or at an outside laboratory.

On Day 1 of Cycle 4, you will have another study visit. You will have all of the same tests performed as you did at the study visits on Day 1 of Cycles 1, 2, and 3. You will also have a bone marrow aspirate and biopsy in order to check the status of the disease. If your bone marrow sample collected at the time of screening showed that you have a mutation in a certain gene, the bone marrow sample collected at this time will be studied further (for a routine test). If this test result shows that the disease has not responded by this time, you will be taken off study.

If the disease has responded by Day 1 of Cycle 4 (or if certain signs and symptoms related to SM have improved), you will continue taking RAD001 for as long as you are benefitting. You will continue having blood (about 2 tablespoons) drawn for routine tests every other week. You will also continue having study visits (with the same tests performed as on Day 1 of Cycle 4), but the visits will be once every 3 months. In other words, you will return on Day 1 of Cycles 4, 7, 10, and so on. On Day 1 of the months when you do not have study visits (Cycles 5, 6, 8, 9, and so on), you will be called on the telephone by the research staff. During these phone calls, you will be asked about any side effects you may have had. You will also be asked about the results of the study-related blood tests that you have had since the last phone call or study visit.

If the disease gets worse, you begin another therapy for cancer, or intolerable side effects occur, you will be taken off study.

This is an investigational study. RAD001 is not Food and Drug Administration (FDA) approved or commercially available. It has been authorized for use in research only. Up to 25 patients will take part in this study. All will be enrolled at M.D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with SM; including mast cell leukemia.
2. Age >/= 18 years
3. Minimum of two weeks since any major surgery or completion of radiation.
4. Eastern Cooperative Oncology Group (ECOG) performance status </= 2
5. Adequate liver function as shown by serum bilirubin </= 1.5 x upper limit of normal (ULN), and serum Alanine transaminase (ALT) </= 3 x ULN
6. Prothrombin Time (PT)/Partial thromboplastin time (PTT)/International normalized ratio (INR) within normal institutional limits
7. Signed informed consent

Exclusion Criteria:

1. Treatment with any conventional (specifically, interferon or cladribine) or investigational medicine for SM within the preceding 4 weeks
2. Chronic treatment with systemic steroids or another immunosuppressive agent
3. Other malignancies within the past 3 years except for adequately treated carcinoma of the cervix or basal or squamous cell carcinomas of the skin, unless patient has SM-associated clonal hematologic disease that does not require therapy, as judged by treating physician and approved by principal investigator.
4. Other concurrent severe and/or uncontrolled medical disease which could compromise participation in the study as judged by the Principal Investigator (i.e., severely impaired lung function, uncontrolled diabetes, uncontrolled hypertension, severe infection, severe malnutrition, unstable angina, or congestive heart failure - New York Heart Association Class III or IV, ventricular arrhythmias, active ischemic heart disease, myocardial infarction within six months, chronic liver or renal disease, active upper GI tract ulceration)
5. A known history of Human immunodeficiency virus (HIV) seropositivity
6. Impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of RAD001 as judged by the Principal Investigator (e.g., ulcerative disease; uncontrolled nausea, vomiting or diarrhea; malabsorption syndrome or small bowel resection)
7. Patients with a bleeding diathesis or on oral anti-vitamin K medication
8. Women who are pregnant or breast feeding, or women/men able to conceive and unwilling to practice an effective method of birth control (women of childbearing potential must have a negative urine or serum pregnancy test within 48 hours prior to administration of RAD001; protocol definition of post-menopausal women is: 12 months of natural (spontaneous) amenorrhea or 6 months of spontaneous amenorrhea with serum FSH levels > 40 mIU/m or 6 weeks post-surgical bilateral oophorectomy with or without hysterectomy)
9. Patients who have received prior treatment with an mTOR inhibitor (e.g., sirolimus, temsirolimus)
10. Patients with a known hypersensitivity to RAD001 (everolimus) or other rapamycins (sirolimus, temsirolimus) or to its excipients
11. Patients unwilling to or unable to comply with the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2007-04; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Srdan Verstovsek, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- The University of Texas M.D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M.D. Anderson's website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period 4/11/2007 to 4/15/2009. All patients registered at The University of Texas M.D. Anderson Cancer Center.
Groups:
- RAD001: Oral RAD001 10 mg daily for 30 days
Period: Overall Study
Arm/Group | RAD001
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | RAD001
Number analyzed (Participants) | 10
Age, Continuous [Median (Full Range); unit: years] | 56 [43 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 4
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Objective Response
Description: Efficacy reported as objective response. Objective response defined as change in serum tryptase level or bone marrow mast cell percentage.
Time Frame: Monthly for first 3 months, then every 3 months
Population: Analysis was per protocol.
Measure: Number; unit: Participants
Arm/Group | RAD001
Number analyzed (Participants) | 10
Participants | 0

ADVERSE EVENTS:
Time Frame: 3 years 7 months
Arm/Group | RAD001
Serious Adverse Events (participants affected / at risk) | 2/10
Other Adverse Events (participants affected / at risk) | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RAD001 (N=10)
Nausea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RAD001 (N=10)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 4 (4)
Mucositis (Gastrointestinal disorders) | 7 (7)
Fatigue (General disorders) | 5 (5)
Fever (General disorders) | 1 (1)
Headache (Nervous system disorders) | 4 (4)
Nausea (Gastrointestinal disorders) | 3 (3)
Vomiting (Gastrointestinal disorders) | 1 (1)
Hyperglycemia (Blood and lymphatic system disorders) | 1 (1)
Hyperlipidemia (Blood and lymphatic system disorders) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes